CLINICAL TRIAL: NCT02037828
Title: The Screening and Confirmation of Protein Markers Which Can Predict the Decline of Lung Function of Chinese Adults in EBC (Exhaled Breathing Condensate )
Brief Title: Exhaled Breathing Condensate (EBC) Features and Lung Function Decline in Chinese Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Guangfa Wang, Pro., Peking University First Hospital
Other Study IDs: PUCRP201303
Record Dates: First submitted 2013-12-25; First posted 2014-01-16 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; biomarker; EBC; FEV1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. EBC
  2. Peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Stable COPD in STEP1: no intervention
- Control in STEP 1: no intervention
- Case group in STEP 2: no intervention
- Control group in STEP2: no intervention

SUMMARY:
Chronic obstructive lung disease (COPD) is a worldwide leading and still increasing cause of chronic morbidity and mortality. The important issue of COPD is its delayed diagnosis. Previous studies have found that accelerated loss of forced expiratory volume in 1 second (FEV1.0) in an individual is considered an indicator of developing COPD. This functional predictive system, due to lower sensitivity, is very difficult to discover high-risk population and earlier stage of the disease. The inflammation occurs earlier than the lung function impairment. Therefore, early detection of the inflammation may theoretically predict the occurrence of COPD and thus may guide early intervention.

Proteomics techniques and protein chip techniques provides us high throughput screening method to figure out characteristic inflammatory or metabolic markers of a diseases. It can be used for searching the biomarkers relating to lung function loss. EBC is collected from exhaled gas and is a good non-invasive method for exploring the pathologic process of the airways.

Thus we designed this study to identify potential biomarkers associated with rapid lung function decline. This study is divided into two parts: 1) screening potential biomarkers between stable COPD and healthy individuals; 2) verifying significant biomarkers of first part in a community-based nested case-control population for 2 years.

DETAILED DESCRIPTION:
Thus we designed this study. This study is divided into two parts: screening target biomarkers and identifying biomarkers.

1. The FIRST STEP is a Case-control study to find target biomarkers. 20 COPD patients and 20 controls are to be enrolled in the study and their EBC and blood are collected. Proteomics techniques and protein chip techniques are to be used to screen COPD specific biomarkers in EBC.
2. The SECOND STEP is a community-based nested case-control study to make sure whether the significant biomarkers in first part can predict rapid decline of lung function. The study will be a community based, multicenter prospective cohort designed, which including a total of 2,400 study subjects. EBC and blood are collected at the baseline and followed up for two years. Case group is defined as subjects with rapid decline of lung function and new COPD patients. Control group is selected according to 1:1 matching with age and gender.

ELIGIBILITY:
1. FIRST STEP:

1. Case Group:

   Inclusion criteria
   1. age from 40 to 75 year olds; gender is not limited.
   2. Stable COPD
   3. Sign the informed consent with willingness of obeying the protocol. Exclusion criteria

   <!-- -->

   1. with known other chronic respiratory diseases except COPD (such as asthma, tuberculosis, bronchiectasis, interstitial lung disease, occupational lung diseases, sarcoidosis, lung cancer, et al);
   2. had been accepted lung lobectomy or transplantation;
   3. be ill with severe, or uncontrolled systemic diseases other than COPD (such as psychiatry diseases, chronic liver diseases, heart failure, auto-immunity diseases, chronic renal diseases, et al );
   4. Alcoholism, drug or solvents addition;
   5. Acute exacerbation COPD patients (AECOPD)
2. Control group:

Inclusion criteria According to age (+ / - 5 years), gender and smoking, to match healthy volunteers as the control group.

1. age from 40 to 75 year olds; gender is not limited.
2. FEV1 /forced vital capacity (FVC)> 70% after inhaling bronchodilators;
3. Sign the informed consent with willingness of obeying the protocol. Exclusion criteria

a. with known other chronic respiratory diseases except COPD (such as asthma, tuberculosis, bronchiectasis, interstitial lung disease, occupational lung diseases, sarcoidosis, lung cancer, et al); b. had been accepted lung lobectomy or transplantation; c. be ill with severe, or uncontrolled systemic diseases other than COPD (such as psychiatry diseases, chronic liver diseases, heart failure, auto-immunity diseases, chronic renal diseases, et al ); d. Alcoholism, drug or solvents addition; e. Acute respiratory infection in 4 weeks (rhinitis, pharyngitis, acute tracheobronchitis, pneumonia, etc.)

2.SECOND STEP: nested case-control study Inclusion criteria

1. age from 40 to 75 year olds; gender is not limited.
2. have been living in the community for more than 1 years and no plan to move in the near 3 years
3. FEV1 / FVC > 70% after inhaling bronchodilators;
4. Sign the informed consent with willingness of obeying the protocol.

Exclusion criteria

1. with known other chronic respiratory diseases except COPD (such as asthma, tuberculosis, bronchiectasis, interstitial lung disease, occupational lung diseases, sarcoidosis, lung cancer, et al);
2. had been accepted lung lobectomy or transplantation;
3. be ill with severe, or uncontrolled systemic diseases other than COPD (such as psychiatry diseases, chronic liver diseases, heart failure, auto-immunity diseases, chronic renal diseases, et al );
4. Alcoholism, drug or solvents addition;

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The FIRST STEP of study will be a outpatient based case-control study. 20 stable COPD patients and 20 healthy individuals will be recruited.
  The SECOND STEP of study will be a community based, multi-center，prospective nested case-control designed, which including a total of 24OO study subjects, it will focus on two different communities, which are Shi Cha Hai community, De Sheng Community in Beijing
Sampling Method: Probability Sample
Enrollment: 2440 (Estimated)
Dates: Start 2014-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Protein biomarkers in EBC predicting rapid decline of lung function | 4 years
  The study(second part) is to identify the biomarkers screened from the first step and make sure which is associated with rapid decline of lung function. The study will be a community based, multicenter prospective cohort designed, which including a total of 2,400 study subjects.

SECONDARY OUTCOMES:
Protein biomarkers of EBC between COPD patients and healthy individuals | 1 year
  The first part of study is to screen target biomarkers. 20 COPD patients and 20 controls are to be enrolled in the study and their EBC are to reserved. Proteomics techniques and protein chip techniques were used to screening COPD specific biomarkers.
Blood biomarkers between COPD patients and healthy individuals | 1 year
  Peripheral blood will be collected. Plasma and PBMC will be extracted and stored respectively.
Blood biomarkers predicting rapid decline of lung function | 4 year
  Peripheral blood will be collected. Plasma and PBMC will be extracted and stored respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Guangfa Wang, MD, PHD, Principal Investigator — Peking Universtiy First Hospital
Locations (1):
- Peking Universtiy First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided